CLINICAL TRIAL: NCT01024673
Title: Clinical Characteristics and Outcomes in Patients Diagnosed With Novel Influenza A (H1N1)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Fernanda P Silveira, MD, MS, MD, University of Pittsburgh
Other Study IDs: IRB#: PRO09090326
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Influenza
Keywords: H1N1
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All the biologic samples and data will be under the control of the principal investigator . To protect confidentiality, all personal identifiers will be removed and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators will keep the samples and data indefinitely. All samples will be stored in the principal investigators laboratory in Scaife Hall, Room 835.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with H1N1: patients who are clinical found to be positive for H1N1 will be enrolled

SUMMARY:
This is study where medical record information will be collected as well as collection of excess biological samples.

DETAILED DESCRIPTION:
Patients diagnosed with H1N1 will be asked to consent and allow us to collect the following:

From the medical record the research staff will review and record the results of the test/procedures (x-rays, CT-scans, EKG (electrocardiogram), etc.) that are part of the subjects clinical care and the results will become part of the research record. We will also collect and record vitals signs, including temperature, blood pressure, heart rate, respiratory rate and record the list of medications the subject is taking. We will also collect information on demographics (address, phone number, etc.) including gender, race and ethnicity, review and record past medical history and any non medical procedures that the subject may have had within the past two months. This information will be collected by the research coordinator from the medical record.

The clinical physician ordered a nasopharyngeal swab or obtained bronchoalveolar lavage fluid to diagnose novel Influenza A (H1N1). We will collect this swab or fluid after the diagnosis has been made, to evaluate the genetic material of the virus. This swab or fluid is normally discarded once the diagnosis is made.

collection of data will be done by the research staff and should not take any longer than 15-20 minutes. The clinical samples that would have been discarded will be collected by the research staff from microbiology and pathology and delivered to the research lab in Scaife.

The investigators will do a 6 month follow up phone call to check the health status of the participant. This will be done by the research coordinator and take no more than 5-10 minutes of the subject's time.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with H1N1

Exclusion Criteria:

* does not meet entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed clinically with H1N1
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-10-15 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
To describe the clinical characteristic and outcomes of the patients admitted to UPMC Presbyterian campus with infection due to novel influenza A (H1N1). | 5 year

SECONDARY OUTCOMES:
To identify risk factors for admission to the ICU and mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silveira, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States